CLINICAL TRIAL: NCT07287553
Title: The Relationship Between Dietary Inflammatory Index and Periodontal Status in Obese Patients
Brief Title: Dietary Inflammatory Index and Periodontal Status in Obese Patients
Status: Recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hatice Yemenoğlu, Doctor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: RecepTayyip ErdoganUniversity
Record Dates: First submitted 2025-11-17; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: obesity; periodontal status; dietary inflammatory index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- anti-inflammatory diet group 1: Individuals on an anti-inflammatory diet
  Interventions: Other: Periodontal indices will be obtained; Other: serum and crevicular fluid samples will be collected
- anti-inflammatory diet group 2: Individuals on an anti-inflammatory diet
  Interventions: Other: Periodontal indices will be obtained; Other: serum and crevicular fluid samples will be collected
- pro-inflammatory diet group 1: individuals on a pro-inflammatory diet
  Interventions: Other: Periodontal indices will be obtained; Other: serum and crevicular fluid samples will be collected
- pro-inflammatory diet group 2: individuals on a pro-inflammatory diet
  Interventions: Other: Periodontal indices will be obtained; Other: serum and crevicular fluid samples will be collected

INTERVENTIONS:
Other: Periodontal indices will be obtained — Periodontal indices will be obtained from all participants
Other: serum and crevicular fluid samples will be collected — Serum and gingival crevicular fluid samples will be collected from all participants.

SUMMARY:
In this study aimed to investigate the effect of nutrition on periodontal status in individuals diagnosed with obesity and without any other systemic disease, and to investigate the relationship between DII and periodontal disease risk. A total of 200 participants will be included in the study. Participants' overall daily Dietary Inflammatory Index (DII) scores will be calculated. The obtained scores will be divided into four groups, from low to high: Q1 (n=50), Q2 (n=50), Q3 (n=50), and Q4 (n=50). According to the DII, groups Q1 and Q2, which include lower scores, represent individuals on an anti-inflammatory diet, while groups Q3 and Q4, which include higher scores, represent individuals on a pro-inflammatory diet. Interleukin (IL)-1β, IL-10, total oxidant status (TOS), and total antioxidant status (TAS) were collected from gingival crevicular fluid (GCF) and serum samples. The levels of biomarkers such as malondialdehyde (MDA), glutathione (GSH), leptin, adiponectin, tumor necrosis factor (TNF)-α and C-reactive protein (CRP) from serum samples alone will be analyzed by ELISA method at the Recep Tayyip Erdoğan University Medical Biochemistry Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with obesity,
* Not having any systemic conditions other than obesity (systemic diseases that may affect periodontal health, such as cardiovascular disease, chronic kidney disease, Type 1 diabetes, Type 2 diabetes, and hypertension (>130/85 mmHg)),
* Being between the ages of 18 and 65,
* Not smoking or consuming alcohol,
* Not having used anti-inflammatory medications in the last 3 months, or antibiotics or systemic corticosteroids in the last 6 months,
* Not being pregnant or lactating,
* Not having received periodontal treatment in the last 6 months,
* Not having received nutritional advice in the last 3 months,
* Obesity diagnosis: BMI > 30 kg/m2 or waist circumference: > 100 cm for men and > 90 cm for women.

Exclusion Criteria:

* Non-obese
* Having any systemic disease other than obesity (such as cardiovascular disease, chronic kidney disease, Type 1 diabetes, Type 2 diabetes, and hypertension (>130/85 mmHg) that may affect periodontal health)
* Being over 65 years old and under 18 years old
* Smoking and alcohol use
* Having used anti-inflammatory drugs in the last 3 months, antibiotics, or systemic corticosteroids in the last 6 months
* Being pregnant or lactating
* Having received periodontal treatment in the last 6 months
* Having received nutritional advice in the last 3 months

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recep Tayyip Erdoğan University
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Periodontal pocket depth | baseline
  The distance between the pocket base and the gingival margin will be measured. It will be measured from the six surfaces of each tooth and the average will be taken higher scores indicate worse outcome.
Clinical attachment loss | baseline
  It will be calculated by measuring the distance between the cementoenemal border and the pocket base. It will be measured from the six surfaces of each tooth and the average will be taken higher scores indicate worse outcome.

SECONDARY OUTCOMES:
interleukin (IL)-1β level | baseline
  IL-1β levels will be measured with biochemical kits.
interleukin (IL)-10 level | baseline
  IL-10 levels will be measured with biochemical kits.
total oxidant status (TOS) level | baseline
  TOS levels will be measured with biochemical kits.
total antioxidant status (TAS) level | baseline
  TAS levels will be measured with biochemical kits.
serum leptin level | baseline
  Leptin levels in serum will be measured with biochemical kits.
serum tumor necrosis factor (TNF)-α level | baseline
  TNF-α levels in serum will be measured with biochemical kits.
serum adiponectin level | baseline
  Adiponectin levels in serum will be measured with biochemical kits.
serum C-reactive protein (CRP) level | baseline
  CRP levels in serum will be measured with biochemical kits.
serum malondialdehyde (MDA) level | baseline
  MDA levels in serum will be measured with biochemical kits.
serum glutathione (GSH) level | baseline
  GSH levels in serum will be measured with biochemical kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University, Rize, Turkey (Türkiye)